CLINICAL TRIAL: NCT03101969
Title: Targeted Intervention (a Telephone Call in the Dominant Language) to Increase Attendance at Scheduled Appointment in an Inner City Academic Pain Clinic
Brief Title: Human Outreach to Improve Adherence With Scheduled Pain Clinic Appointments
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Michael Andreae, Anesthesiologist, Montefiore Medical Center
Other Study IDs: 2014-3683
Record Dates: First submitted 2016-06-29; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Patient Compliance
Keywords: language; scheduled; appointment
MeSH Terms: conditions — Patient Compliance; Language | interventions — CD56 Antigen

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Call — not called, not reached, and spoken to

SUMMARY:
Patients tend to miss their scheduled appointments in chronic pain clinics for unknown reasons. This study will test the hypothesis in a prospective pragmatic trial that a human telephone call in the primary language of the patient, promising a clinical encounter in this language improves attendance at scheduled appointments in an academic inner city pain clinic.

DETAILED DESCRIPTION:
Language barriers may lead to poor attendance at pain clinic appointments, especially in underserved patients. Targeted interventions can help overcome barriers and significantly improve adherence, but have rarely been rigorously investigated in randomized clinical trials. Our objective is to investigate if (1) making a telephone call in the patient's preferred language increases adherance with scheduled appointment in an inner city academic pain clinic or at least reduces failure to attend without a prior cancellation call and (2) if this intervention is more effective in Spanish speakers.

After institutional review board approval and waiver of informed consent, we enroll all adult patients (18 years and up) with a scheduled first appointment at our outpatient Pain Center at Montefiore Medical Center located in the Bronx, New York from October 2014 through October 2015. Participants are randomized to receive a phone call in their preferred language before their appointment, or not. We recorded if participants attended as scheduled and/or called to cancel. We fit stratified and multivariate multinomial logistic regression models.

In a methodologically rigorous randomized design, we seek to demonstrate that a human phone call in the patient's primary language increases adherence with scheduled appointments in an ethnically diverse, poor population, typical for an inner city pain clinic. Our targeted intervention may provide considerable cost savings to the institution while bolstering the patient-doctor relationship and overcoming barriers to access much needed care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have scheduled appointment at Montefiore Medical Center

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are 18 years of age and older that has a scheduled appointment at Montefiore Medical Center.
Sampling Method: Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Patient attendance at scheduled pain clinic appointment | 1day
  patient attends a scheduled appointment at a chronic pain clinic the day after the call or not, as ascertained from the clinic attendance sheet

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes